CLINICAL TRIAL: NCT03346733
Title: The Effect of Psyllium Fibre (Plantago Ovata) on LDL-cholesterol and Emerging Lipid Targets, Non-HDL-cholesterol and Apolioprotein-B: A Systematic Review and Meta-analysis of Randomized Controlled Trials
Brief Title: The Effect of Psyllium Fibre on LDL-C, Non-HDL-C, and Apolioprotein-B: A Systematic Review and Meta-analysis
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Unity Health Toronto (Other)
Responsible Party: Sponsor
Other Study IDs: Psyllium_Chol SR&MA
Record Dates: First submitted 2017-11-15; First posted 2017-11-17 (Actual); Last update posted 2017-11-17 (Actual); Status verified 2017-11

CONDITIONS: Hypercholesterolemia; Cardiovascular Risk Factor
Keywords: psyllium; viscous fibre
MeSH Terms: conditions — Hypercholesterolemia

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Dietary Supplement: Psyllium Fibre — Viscous soluble psyllium fibre

SUMMARY:
Serum cholesterol is a major modifiable risk factor for cardiovascular disease, which despite considerable reduction in prevalence, remains the leading cause of premature mortality worldwide. Although LDL-C continues to be recognized as the primary therapeutic target, accumulating evidence suggests that alternative lipid parameters, non-HDL-C and apoB, may provide predictive value beyond that of LDL-C alone, in most population categories. Numerous lifestyle strategies have been developed to manage elevated cholesterol concentrations, of which viscous fibre is often encouraged for its beneficial effects on LDL-C reduction. Conversely, the effects of viscous fibre on new lipid markers, non-HDL and apoB, have yet to be defined. Therefore, this study seeks to elucidate the therapeutic potential of psyllium fibre on totality of atherogenic cholesterol and lipoprotein particles in a systematic review and meta-analysis of randomized controlled trials.

DETAILED DESCRIPTION:
Background: Studies have identified viscous dietary fibre as potentially attenuating cholesterol, including psyllium husk that reduces LDL-cholesterol (LDL-C) thus, may alleviate cardiovascular disease (CVD) treatment.

Objective: To update evidence on the effect of psyllium on LDL-C, and provide assessment of its impact on new lipid markers: non-HDL cholesterol (non-HDL-C) and apolipoprotein-B (apoB).

Design: Conduct of the systematic review and meta-analysis will follow the Cochrane handbook for systematic reviews of interventions. The reporting will follow the Preferred Reporting Items for Systematic reviews and Meta-Analyses (PRISMA) guidelines.

Data Sources & Study Selection: MEDLINE, EMBASE, CINAHL and The Cochrane Central Register of Controlled Trials will be searched using appropriate search terms. Independent reviewers will extract information about study design, sample size, subject characteristics, dose, follow-up, and placebo/compare. RCTs that investigate the effect of psyllium fibre on LDL-C, non-HDL-C or apoB will be included with a minimum follow-up period ≥ 3 weeks. The amount of psyllium fibre must be reported and effects on outcomes LDL-C, non-HDL-C or apoB must be isolatable. Studies detailing sufficient information for non-HDL-C calculation will also be considered. Unpublished trials are considered and no restriction placed on language.

Outcomes: LDL-C, non-HDL-C, apoB

Data Extraction: Mean±SEM values will be extracted for all outcomes. Standard computations and imputations will be used to derive missing variance data. Risk of bias and overall study quality will be assessed using the Cochrane Risk of Bias tool and GRADE approach.

Data Synthesis: Data will be pooled using the generic inverse variance method with random effects models. Heterogeneity assessed by the Cochran Q-statistic and quantified by I2. Sensitivity analysis and a priori subgroup analyses will be performed to explore sources of heterogeneity. A spline curve model (MKSPLINE procedure) will be utilized to illustrate a non-linear dose-response curve. Publication bias will be investigated by visual inspection of funnel plots and formally tested using Egger's and Begg's tests. If significant, a Trim and Fill analyses will be performed.

ELIGIBILITY:
Inclusion Criteria:

* human trials
* RCT that investigates the effect of psyllium fibre on LDL-C, non-HDL-C and/or apoB
* suitable control
* minimum follow up period ≥ 3 weeks
* amount of psyllium fibre must be report and effect on outcomes isolatable

Exclusion Criteria:

* follow up < 3 weeks
* non-human trials
* lack of suitable control
* no viable endpoint data

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Hypercholesterolemic or normocholesterolemic children and adults, overweight and obese individuals or individuals with diabetes
Sampling Method: Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2013-10-08 (Actual); Primary Completion 2017-11 (Estimated); Study Completion 2017-12 (Estimated)

PRIMARY OUTCOMES:
LDL-Cholesterol | >= 3 months
non-HDL cholesterol | >= 3 months
Apolipoprotein-B | >= 3 months

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Jovanovski E, Yashpal S, Komishon A, Zurbau A, Blanco Mejia S, Ho HVT, Li D, Sievenpiper J, Duvnjak L, Vuksan V. Effect of psyllium (Plantago ovata) fiber on LDL cholesterol and alternative lipid targets, non-HDL cholesterol and apolipoprotein B: a systematic review and meta-analysis of randomized controlled trials. Am J Clin Nutr. 2018 Nov 1;108(5):922-932. doi: 10.1093/ajcn/nqy115. PMID 30239559